CLINICAL TRIAL: NCT03797742
Title: A Clinical Follow-up Study of Heart Failure Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HF201801
Record Dates: First submitted 2019-01-01; First posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum; Whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NC: Patients without heart failure.
- DCM: Dilated cardiomyopathy patients.
- ICM: Ischemic cardiomyopathy patients.

SUMMARY:
Heart failure (HF), a current worldwide pandemic with an unacceptable high level of morbidity and mortality, brings an enormous medical and societal burden. Chronic HF is characterized by progressive alteration of cardiac structure and function. But the molecular mechanism of these alterations is still not well-established and needs to be discussed further. HF is a highly heterogeneous disease that can be caused by a multiple of diseases. Dilated cardiomyopathy (DCM) and ischemic cardiomyopathy (ICM) are the main causes of this syndrome. Although HF is the common manifestation of DCM and ICM, the etiology and pathogenesis are different. Understanding the different pathophysiological mechanisms will contribute to the prevention and individualized therapy of heart failure. Therefore, this study aims to observation the different characteristics of the molecular biology and clinical courses in DCM and ICM patients.

ELIGIBILITY:
Inclusion Criteria:

* LVEF≤ 55%
* enlarged left ventricular end-diastolic dimension
* ICM group: with history of MI or revascularization; ≥ 75% stenosis of LM or proximal LAD; ≥ 75% stenosis of two or more epicardial vessels.
* symptomatic heart failure

Exclusion Criteria:

* Known malignant tumour diseases
* Pregnancy or lactation period；
* Investigators think not suitable to participate in this trial.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The inpatient in the department of cardiology of Zhongshan Hospital, Fudan University will be selected.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
NYHA functional class | one year after enrolled
  NYHA cardiac functional class
All-cause mortality | one year after enrolled
  All-cause mortality during follow-up

SECONDARY OUTCOMES:
hospitalization for cardiac causes | one year after enrolled
  hospitalization for cardiac causes during follow-up
left ventricular end-diastolic dimension(LVEDD) dilates. | one year after enrolled
  left ventricular structure changes:left ventricular end-diastolic dimension(LVEDD) dilates.
left ventricular ejection fraction reduces | one year after enrolled
  left ventricular function changes:left ventricular ejection fraction reduces

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, China